CLINICAL TRIAL: NCT00005858
Title: Phase I Study of LMB-9, a Recombinant Disulfide Stabilized Anti-Lewis Y Immunotoxin Admistered by Continuous Infusion
Brief Title: LMB-9 Immunotoxin in Treating Patients With Advanced Colon, Breast, Non-small Cell Lung, Bladder, Pancreatic, or Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSGCC-9981; CDR0000067885 (Registry Identifier: PDQ (Physician Data Query)); MSGCC-IRB-0200123; NCI-511
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Bladder Cancer; Breast Cancer; Colorectal Cancer; Lung Cancer; Ovarian Cancer; Pancreatic Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; recurrent non-small cell lung cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; recurrent colon cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; ovarian stromal cancer; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; male breast cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Breast Neoplasms, Male

ARMS (1):
- Arm I (Experimental): Patients receive LMB-9 immunotoxin IV continuously for 10 days. Treatment continues every 30 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of LMB-9 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Biological: LMB-9 immunotoxin

INTERVENTIONS:
Biological: LMB-9 immunotoxin

SUMMARY:
Phase I trial to study the effectiveness of LMB-9 immunotoxin in treating patients who have advanced colon, breast, non-small cell lung, bladder, pancreatic, or ovarian cancer. The LMB-9 immunotoxin can locate tumor cells and kill them without harming normal cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of LMB-9 immunotoxin in patients with advanced colon, breast, non-small cell lung, bladder, pancreas, or ovarian cancer.

II. Assess the toxicity and pharmacokinetics of this treatment regimen in these patients.

III. Determine the clinical responses in patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients receive LMB-9 immunotoxin IV continuously for 10 days. Treatment continues every 30 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of LMB-9 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 weeks and then every 2 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced colon, breast, non-small cell lung, bladder, pancreas, or ovarian cancer refractory to standard treatment or for which no effective standard therapy exists
* Expresses Lewis Y antigen
* Evidence of disease progression
* B3 antigen on the surface of more than 30% of the tumor cells determined by immunohistochemistry
* No neutralizing antibodies to LMB-9 immunotoxin
* No untreated CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Performance status:

* ECOG 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute granulocyte count greater than 1,200/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT and SGPT no greater than 2.5 times upper limit of normal (liver metastases allowed)
* Albumin at least 3.0 g/dL
* No prior liver disease (e.g., alcohol liver disease)
* Hepatitis B and C negative

Renal:

* Creatinine no greater than 1.4 mg/dL
* Creatinine clearance greater than 60 mL/min
* Proteinuria less than 1 g/24 hours

Cardiovascular:

* No history of coronary artery disease
* No cardiac arrhythmia requiring therapy
* No New York Heart Association class II-IV congestive heart failure

Pulmonary:

* Pulmonary function test required if significant smoking history, possible pulmonary disease, or lung cancer
* FEV1 and FVC at least 65% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known seizure disorders
* No urinary tract infection
* No other concurrent malignancy
* No active peptic ulcer disease
* No known allergy to omeprazole
* No contraindication to pressor therapy
* No other concurrent medical or psychological condition that would preclude study

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered

Endocrine therapy:

* At least 3 weeks since prior hormonal therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2000-04 (Actual); Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith E. Karp, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland